CLINICAL TRIAL: NCT06083051
Title: Randomized Clinical Trial Evaluating Differences in Postoperative Symptoms With 6Fr Percuflex Ureteral Stents Versus 6Fr Tria Ureteral Stents Versus 4.8Fr Percuflex Ureteral Stents Versus 4.8Fr Tria Ureteral Stents After Laser Lithotripsy of Renal and Ureteral Stones
Brief Title: Differences in Postoperative Symptoms With Four Ureteral Stents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-0832; Urology (Other: UW Madison); Protocol Version 10/28/2024 (Other: UW Madison)
Record Dates: First submitted 2023-10-09; First posted 2023-10-13 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Urinary Stone
MeSH Terms: conditions — Urinary Calculi

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- 6Fr Percuflex ureteral stents (Active Comparator)
  Interventions: Device: 6Fr Percuflex ureteral stents
- 6Fr Tria ureteral stents (Active Comparator)
  Interventions: Device: 6Fr Tria ureteral stents
- 4.8Fr Tria ureteral stents (Active Comparator)
  Interventions: Device: 4.8Fr Tria ureteral stents
- 4.8Fr Percuflex ureteral stents (Active Comparator)
  Interventions: Device: 4.8Fr Percuflex ureteral stents

INTERVENTIONS:
Device: 6Fr Percuflex ureteral stents — The Percuflex stent is a 6Fr polymeric, hydrophilic coated stent that is routinely used post ureteroscopy with laser lithotripsy.
  Arms: 6Fr Percuflex ureteral stents
Device: 6Fr Tria ureteral stents — The Tria stent is a new stent that is designed to soften at body temperature after placement, with an additional coating that prevents calcium and magnesium build up. This is intended to increase patient tolerability of the stent. 6 Fr is the diameter.
  Arms: 6Fr Tria ureteral stents
Device: 4.8Fr Tria ureteral stents — The Tria stent is a new stent that is designed to soften at body temperature after placement, with an additional coating that prevents calcium and magnesium build up. This is intended to increase patient tolerability of the stent. 4.8 Fr is the diameter.
  Arms: 4.8Fr Tria ureteral stents
Device: 4.8Fr Percuflex ureteral stents — The Percuflex stent is a 4.8Fr polymeric, hydrophilic coated stent that is routinely used post ureteroscopy with laser lithotripsy.
  Arms: 4.8Fr Percuflex ureteral stents

SUMMARY:
This is a prospective randomized controlled trial designed to assess the differences in postoperative symptoms related to placement of a 6Fr Percuflex ureteral stents, 6Fr Tria ureteral stents, 4.8Fr Percuflex ureteral stents, and 4.8Fr Tria ureteral stents after ureteroscopy with laser lithotripsy for treatment of upper tract urinary stones. 272 participants will be enrolled and will be on study for up to approximately 10 weeks.

DETAILED DESCRIPTION:
The investigators will compare Ureteral Stent Symptom Questionnaire (USSQ) scores with each ureteral stent. Laser lithotripsy is a surgical procedure performed during stone surgeries. The Percuflex ureteral stent and Tria ureteral stent are FDA approved and clinically used in the United States.

A total of 3 clinic visits (i.e., pre-operative visit, the stent removal 1-2 weeks after surgery, and one post-operative visit 3-6 weeks after surgery) in addition to the surgery will be needed for this study. The patient's demographic information and medical background data will be collected from the medical record.

The USSQ will be administered twice:

1. At the time of stent removal (1-2 weeks after surgery ) (This is standard of care)
2. At the first postoperative follow-up after stent removal (3-6 weeks) (This is the standard of care).

The following information will be collected as secondary outcomes:

1. WisQOL which will be administered three times. It is UW standard of care for stone patients to complete the WisQOL at every clinic visit.
2. ER visits documented in patients chart
3. Unscheduled clinic follow-up documented in patient chart
4. Additional prescriptions for stent related symptoms documented by patient chart
5. Stent complications by fluoroscopy or image
6. Physician evaluation of the stent. Physicians will complete a one page survey at the end of the case evaluating the stent.

ELIGIBILITY:
Inclusion Criteria:

* Patients with renal or ureteral urinary stones who require endoscopic treatment and stent placement in the outpatient operating room.

Exclusion Criteria:

* Pregnant patients
* Patients with transplant kidneys
* Patients with irreversible coagulopathy
* Patients with known ureteral stricture disease
* Non-English speaking, vulnerable patients such as lacking of decision-making capability, prisoner, adult unable to consent, will not be enrolled.
* Patients with planned staged procedures.
* Patients who have stent placed before surgery.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Start 2024-03-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Ureteral Stent Symptom Questionnaire (USSQ) scores-Urinary symptoms | at time of stent removal 1-2 weeks after surgery (up to 4 weeks on study)
  USSQ is a 38-item questionnaire to evaluate symptoms and impact on quality of life of ureteral stents. The high scores indicate worse outcomes. It has 5 sections, urinary symptoms, pain, general health, work performance, and sexual matters. The urinary subscale score range from 11-54.
Ureteral Stent Symptom Questionnaire (USSQ) scores-Pain Index | at time of stent removal 1-2 weeks after surgery (up to 4 weeks on study)
  USSQ is a 38-item questionnaire to evaluate symptoms and impact on quality of life of ureteral stents. The high scores indicate worse outcomes. It has 5 sections, urinary symptoms, pain, general health, work performance, and sexual matters. The Pain subscale score range from 6-37.
Ureteral Stent Symptom Questionnaire (USSQ) scores-General Health | at time of stent removal 1-2 weeks after surgery (up to 4 weeks on study)
  USSQ is a 38-item questionnaire to evaluate symptoms and impact on quality of life of ureteral stents. The high scores indicate worse outcomes. It has 5 sections, urinary symptoms, pain, general health, work performance, and sexual matters. The General Health subscale score range from 6-28.
Ureteral Stent Symptom Questionnaire (USSQ) scores-Work Performance | at time of stent removal 1-2 weeks after surgery (up to 4 weeks on study)
  USSQ is a 38-item questionnaire to evaluate symptoms and impact on quality of life of ureteral stents. The high scores indicate worse outcomes. It has 5 sections, urinary symptoms, pain, general health, work performance, and sexual matters. The Work Performance subscale score range from 3-15.
Ureteral Stent Symptom Questionnaire (USSQ) scores-Sexual matters | at time of stent removal 1-2 weeks after surgery (up to 4 weeks on study)
  USSQ is a 38-item questionnaire to evaluate symptoms and impact on quality of life of ureteral stents. The high scores indicate worse outcomes. It has 5 sections, urinary symptoms, pain, general health, work performance, and sexual matters. The Sexual Matters subscale score range from 2-10.
Ureteral Stent Symptom Questionnaire (USSQ) scores-Urinary symptoms | at time of stent removal 3-6 weeks after surgery (up to 10 weeks on study)
  USSQ is a 38-item questionnaire to evaluate symptoms and impact on quality of life of ureteral stents. The high scores indicate worse outcomes. It has 5 sections, urinary symptoms, pain, general health, work performance, and sexual matters. The urinary subscale score range from 11-54.
Ureteral Stent Symptom Questionnaire (USSQ) scores-Pain index | at time of stent removal 3-6 weeks after surgery (up to 10 weeks on study)
  USSQ is a 38-item questionnaire to evaluate symptoms and impact on quality of life of ureteral stents. The high scores indicate worse outcomes. It has 5 sections, urinary symptoms, pain, general health, work performance, and sexual matters. The Pain subscale score range from 6-37.
Ureteral Stent Symptom Questionnaire (USSQ) scores-General Health | at time of stent removal 3-6 weeks after surgery (up to 10 weeks on study)
  USSQ is a 38-item questionnaire to evaluate symptoms and impact on quality of life of ureteral stents. The high scores indicate worse outcomes. It has 5 sections, urinary symptoms, pain, general health, work performance, and sexual matters. The Pain subscale score range from 6-28.
Ureteral Stent Symptom Questionnaire (USSQ) scores-Work Performance | at time of stent removal 3-6 weeks after surgery (up to 10 weeks on study)
  USSQ is a 38-item questionnaire to evaluate symptoms and impact on quality of life of ureteral stents. The high scores indicate worse outcomes. It has 5 sections, urinary symptoms, pain, general health, work performance, and sexual matters. The Work Performance subscale score range from 3-15.
Ureteral Stent Symptom Questionnaire (USSQ) scores-Sexual Matters | at time of stent removal 3-6 weeks after surgery (up to 10 weeks on study)
  USSQ is a 38-item questionnaire to evaluate symptoms and impact on quality of life of ureteral stents. The high scores indicate worse outcomes. It has 5 sections, urinary symptoms, pain, general health, work performance, and sexual matters. The Sexual Matters subscale score range from 2-10.

SECONDARY OUTCOMES:
Change in Quality of Life measured by WISQOL Scores | pre-operative visit (baseline), the stent removal 1-2 weeks after surgery (up to 4 weeks on study), and one post-operative visit 3-6 weeks after surgery (up to 10 weeks on study)
  WISQOL short form is a 6 item questionnaire which can be scored from 1 (worst outcome) to 5 (best outcome). The raw score range is 5-30. In the study, standardized total score is used. The range of the standardized total score is 0-100.
Number of Emergency Room Visits | up to 10 weeks
  Data collected from medical record.
Number of Unscheduled Clinic Follow-Ups | up to 10 weeks
  Data collected from medical record.
Summary of Additional Prescriptions for Stent-Related Symptoms | up to 10 weeks
  Data collected from medical record.
Summary of Stent Complications | up to 10 weeks
Physician Evaluation of Stent: Survey Scores | up to 10 weeks
  Physicians will complete a one page survey at the end of the case evaluating the stent. Scores are from 0-5 where higher scores indicate a more positive evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Antar, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No